CLINICAL TRIAL: NCT00487136
Title: Multiple-Dose Pharmacokinetic and Pharmacodynamic Interaction Between ABT-335, Rosuvastatin and Warfarin
Brief Title: Interaction Between ABT-335, Rosuvastatin and Warfarin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Maureen Kelly, MD, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M06-887
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: Drug Interaction; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — Warfarin; 2-(4-(4-chlorobenzoyl)phenoxy)-2-methylpropanoic acid; Rosuvastatin Calcium; fenofibric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Warfarin (Active Comparator): Warfarin fixed dose plus one capsule containing placebo for ABT-335, one placebo tablet to match rosuvastatin 5 mg and one placebo tablet to match rosuvastatin 20 mg, administered for 10 consecutive days.
  Interventions: Drug: Warfarin
- Warfarin plus ABT-335 plus Rosuvastatin (Experimental): Warfarin fixed dose plus one capsule containing ABT-335 mini-tablets equivalent to 135 mg fenofibric acid, one 5 mg tablet of rosuvastatin and one tablet of placebo to match rosuvastatin 20 mg, administered for 10 consecutive days.
  Interventions: Drug: warfarin plus ABT-335 plus rosuvastatin 5 mg
- Warfarin plus ABT-335 mg plus rosuvastatin 20 mg (Experimental): Warfarin fixed dose plus one capsule containing ABT-335 mini-tablets equivalent to 135 mg fenofibric acid, one tablet of placebo to match rosuvastatin 5 mg and one 20 mg tablet of rosuvastatin, administered for 10 consecutive days.
  Interventions: Drug: warfarin plus ABT-335 plus rosuvastatin 20 mg

INTERVENTIONS:
Drug: Warfarin — Warfarin fixed dose plus one capsule containing placebo for ABT-335, one placebo tablet to match rosuvastatin 5 mg and one placebo tablet to match rosuvastatin 20 mg, administered for 10 consecutive days.
  Other Names: Coumadin
  Arms: Warfarin
Drug: warfarin plus ABT-335 plus rosuvastatin 5 mg — Warfarin fixed dose plus one capsule containing ABT-335 mini-tablets equivalent to 135 mg fenofibric acid, one 5 mg tablet of rosuvastatin and one tablet of placebo to match rosuvastatin 20 mg, administered for 10 consecutive days.
  Other Names: warfarin; coumadin ABT-335; fenofibric acid; Trilipix Rosuvastatin; Crestor
  Arms: Warfarin plus ABT-335 plus Rosuvastatin
Drug: warfarin plus ABT-335 plus rosuvastatin 20 mg — Warfarin fixed dose plus one capsule containing ABT-335 mini-tablets equivalent to 135 mg fenofibric acid, one tablet of placebo to match rosuvastatin 5 mg and one 20 mg tablet of rosuvastatin, administered for 10 consecutive days.
  Other Names: warfarin; coumadin; ABT-335; fenofibric acid; Trilipix Rosuvastatin; Crestor
  Arms: Warfarin plus ABT-335 mg plus rosuvastatin 20 mg

SUMMARY:
This is a multiple-dose, double-blind, randomized, single-center, parallel-group study in adult male subjects in general good health.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) is 19 to 29, inclusive.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).
* Written informed consent prior to the initiation of screening or study-specific procedures.

Exclusion Criteria:

* Subjects with unstable medical conditions or medical conditions considered inappropriate in a clinical trial.
* Subjects taking concomitant medications.
* Subjects with a recent history of surgery or trauma.
* Subjects with a history of any bleeding disorder.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2007-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters, pharmacodynamic variables | Day 24

SECONDARY OUTCOMES:
Vital signs, physical examinations, laboratory tests, ECGs, adverse events | Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Torbjörn Lundström, MD, Study Director — AstraZeneca
Locations (1):
- Site Ref # / Investigator 5290, Little Rock, Arkansas, United States